CLINICAL TRIAL: NCT00351390
Title: The Use of Pro-Brain Natriuretic Peptide Targeted Therapy to Tailor Medical Management of Patients With Congestive Heart Failure Followed in an Outpatient Setting: the ProBNP Outpatient Tailored CHF Therapy (PROTECT) Study
Brief Title: Use of NT-proBNP Testing to Guide Heart Failure Therapy in the Outpatient Setting.
Acronym: PROTECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Roche Diagnostics GmbH (Industry)
Responsible Party: Principal Investigator, James L. Januzzi, Dr., Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004-P-001447/12
Record Dates: First submitted 2006-07-10; First posted 2006-07-12 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Congestive Heart Failure
Keywords: congestive heart failure treatment; congestive heart failure, prognosis; NT-proBNP testing
MeSH Terms: conditions — Heart Failure | interventions — Drug Therapy

ARMS (2):
- SOC (Placebo Comparator): Standard of care HF therapy without NT-proBNP guidance
  Interventions: Other: Drug therapy for HF
- NT-proBNP arm (Active Comparator): NT-proBNP plus standard HF management
  Interventions: Other: NT-proBNP guided HF therapy

INTERVENTIONS:
Other: Drug therapy for HF — Titration of HF meds in an aggressive out patient manner following guideline direction
  Arms: SOC
Other: NT-proBNP guided HF therapy — Standard of care drug therapy following guideline direction, plus adjustment of medication titrated to achieve NT-proBNP <1000 pg/mL
  Arms: NT-proBNP arm

SUMMARY:
Levels of amino-terminal pro-brain natriuretic peptide (NT-proBNP) a hormone released from the heart in patients with heart failure (HF) are strongly prognostic of adverse events, such as hospitalization or death from HF. Therapies that are beneficial for HF (such as beta blockers or angiotensin converting enzyme inhibitors) tend to lower levels of NT-proBNP in parallel with improvements in outcomes of patients so treated. Importantly, Nt-proBNP levels may identify a patient at high risk for adverse outcome from their HF, even in periods of apparent stability.

It remains unclear, however, whether treating patients based on their NT-proBNP concentrations would be associated with better outcomes compared to standard HF therapy without measurement of NT-proBNP values.

The goal of the PROTECT study is to evaluate whether treatment of patients with advanced and recently destabilized HF would benefit from NT-proBNP guided HF treatment, compared to standard HF therapy without such 'hormone guided' treatment.

DETAILED DESCRIPTION:
300 patients with class II-IV heart failure (HF) due to systolic dysfunction (left ventricular ejection fraction <40%) and recent (within 6 months) destabilized HF will be randomized 1:1 to either 'standard of care' therapy for their HF versus 'standard of care plus NT-proBNP guided' care.

At randomization, patients at MGH will undergo a 2-dimensional echocardiogram for cardiac structure and function.

Patients randomized to the 'standard of care' arm of the study will receive aggressive therapy for their HF, including evidence-based addition/titration of therapeutic agents in the trial, such as carvedilol or metoprolol XL, angiotensin converting enzyme inhibitors or angiotensin receptor blockers, spironolactone inhibitors (for those in class III or IV), digoxin (when applicable), loop diuretics, as well as nitrates with or without hydralazine. Biventricular pacing with/without ICD capability will be performed at the discretion of the investigator. Any changes in therapy will be accompanied by a 2 week follow up for re-assessment and further titration of medications, based on clinical judgment.

At each interim visit, patients in the 'standard of care' arm will have a Minnesota Living with Heart Failure questionnaire taken. For all visits, including those triggered by med changes, laboratories will be checked including serum chemistries; a sample of blood for blinded NT-proBNP, troponin T, and high sensitivity CRP will be obtained for measurement after the trial is complete.

Patients randomized to the 'standard of care plus NT-proBNP guided' arm will receive the same aggressive medical care as above, but will also have an unblinded measurement of NT-proBNP provided to the study investigator within an hour of first patient contact. Therapeutic decision-making will be first based on clinical acumen/judgment, but if the NT-proBNP is elevated, per protocol, the investigator will adjust therapies accordingly, including escalation of existing therapies with known effects on NT-proBNP levels, as well as possible addition of similar therapies not yet in use (such as spironolactone).

Patients will be followed for events including destabilized HF (in or outpatient), cardiovascular events (including ischemic complications, ICD discharge, or development of non-fatal arrhythmia such as atrial fibrillation), or death.

At the end of one year, event rates will be assessed and the outcomes in the two arms will be compared. As well, echocardiography will be performed on subjects at one year and differences from baseline in both groups will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age > 21 years of age
* Left ventricular ejection fraction ≤ 40%
* NYHA class II-IV heart failure
* Hospital admission, Emergency Department visit, or outpatient diuretic escalation of therapy for destabilized HF at least once in the 6 months prior to enrollment

Exclusion Criteria:

* Severe renal insufficiency defined as serum creatinine > 2.5 mg/dl
* Inoperable aortic valvular heart disease
* Life expectancy <1 year due to causes other than HF such as advanced cancer
* Cardiac transplantation or revascularization indicated or expected within 6 months
* Severe obstructive or restrictive pulmonary disease, defined as a forced expiratory volume in 1S <1 L when diagnosed as standard of care.
* Subject unable or unwilling to provide written informed consent
* Coronary revascularization (PCI or CABG) within the previous 3 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2005-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Effect of Standard of Care therapy versus Standard of Care plus NT-proBNP targeted therapy on total cardiovascular events | One year

SECONDARY OUTCOMES:
Effect of Standard of Care therapy versus Standard of Care plus NT-proBNP targeted therapy on the reduction of outpatient decompensated HF. | One year
Effect of Standard of Care therapy versus Standard of Care plus NT-proBNP targeted therapy on change in NT-proBNP levels, both the change in absolute value as well as in relative value, from baseline to end of study. | One year
Effect of Standard of Care therapy versus Standard of Care plus NT-proBNP targeted therapy alone on echocardiographic parameters including LV systolic and diastolic function, RV systolic and diastolic function, RV systolic pressures, degree of valvular | One year
Effect of Standard of Care therapy versus Standard of Care plus NT-proBNP targeted therapy on the reduction of all cause mortality. | One year
Ability of cTnT and hsCRP, independently as well as together with NT-proBNP, to predict cardiovascular endpoints. | One year
Effect of Standard of Care therapy versus Standard of Care plus NT-proBNP targeted therapy alone on patient quality of life. | One year
Cost benefits of NT-proBNP guided HF therapy versus standard of care. | One year

CONTACTS AND LOCATIONS:
Overall Officials: James L. Januzzi, MD, FACC, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Shah R, Ziegler O, Yeri A, Liu X, Murthy V, Rabideau D, Xiao CY, Hanspers K, Belcher A, Tackett M, Rosenzweig A, Pico AR, Januzzi JL, Das S. MicroRNAs Associated With Reverse Left Ventricular Remodeling in Humans Identify Pathways of Heart Failure Progression. Circ Heart Fail. 2018 Feb;11(2):e004278. doi: 10.1161/CIRCHEARTFAILURE.117.004278. PMID 29438982
- [Derived] Motiwala SR, Gaggin HK, Gandhi PU, Belcher A, Weiner RB, Baggish AL, Szymonifka J, Januzzi JL Jr. Concentrations of highly sensitive cardiac troponin-I predict poor cardiovascular outcomes and adverse remodeling in chronic heart failure. J Cardiovasc Transl Res. 2015 Apr;8(3):164-72. doi: 10.1007/s12265-015-9618-4. Epub 2015 Mar 17. PMID 25777344
- [Derived] Gandhi PU, Motiwala SR, Belcher AM, Gaggin HK, Weiner RB, Baggish AL, Fiuzat M, Brunner-La Rocca HP, Januzzi JL Jr. Galectin-3 and mineralocorticoid receptor antagonist use in patients with chronic heart failure due to left ventricular systolic dysfunction. Am Heart J. 2015 Mar;169(3):404-411.e3. doi: 10.1016/j.ahj.2014.12.012. Epub 2015 Jan 7. PMID 25728731
- [Derived] Gaggin HK, Szymonifka J, Bhardwaj A, Belcher A, De Berardinis B, Motiwala S, Wang TJ, Januzzi JL Jr. Head-to-head comparison of serial soluble ST2, growth differentiation factor-15, and highly-sensitive troponin T measurements in patients with chronic heart failure. JACC Heart Fail. 2014 Feb;2(1):65-72. doi: 10.1016/j.jchf.2013.10.005. Epub 2014 Jan 25. PMID 24622120
- [Derived] Motiwala SR, Szymonifka J, Belcher A, Weiner RB, Baggish AL, Gaggin HK, Bhardwaj A, Januzzi JL Jr. Measurement of novel biomarkers to predict chronic heart failure outcomes and left ventricular remodeling. J Cardiovasc Transl Res. 2014 Mar;7(2):250-61. doi: 10.1007/s12265-013-9522-8. Epub 2013 Dec 6. PMID 24309956
- [Derived] Gaggin HK, Motiwala S, Bhardwaj A, Parks KA, Januzzi JL Jr. Soluble concentrations of the interleukin receptor family member ST2 and beta-blocker therapy in chronic heart failure. Circ Heart Fail. 2013 Nov;6(6):1206-13. doi: 10.1161/CIRCHEARTFAILURE.113.000457. Epub 2013 Oct 10. PMID 24114865
- [Derived] Bhardwaj A, Rehman SU, Mohammed AA, Gaggin HK, Barajas L, Barajas J, Moore SA, Sullivan D, Januzzi JL. Quality of life and chronic heart failure therapy guided by natriuretic peptides: results from the ProBNP Outpatient Tailored Chronic Heart Failure Therapy (PROTECT) study. Am Heart J. 2012 Nov;164(5):793-799.e1. doi: 10.1016/j.ahj.2012.08.015. PMID 23137512
- [Derived] Weiner RB, Baggish AL, Chen-Tournoux A, Marshall JE, Gaggin HK, Bhardwaj A, Mohammed AA, Rehman SU, Barajas L, Barajas J, Gregory SA, Moore SA, Semigran MJ, Januzzi JL Jr. Improvement in structural and functional echocardiographic parameters during chronic heart failure therapy guided by natriuretic peptides: mechanistic insights from the ProBNP Outpatient Tailored Chronic Heart Failure (PROTECT) study. Eur J Heart Fail. 2013 Mar;15(3):342-51. doi: 10.1093/eurjhf/hfs180. Epub 2012 Nov 6. PMID 23132825
- [Derived] Gaggin HK, Mohammed AA, Bhardwaj A, Rehman SU, Gregory SA, Weiner RB, Baggish AL, Moore SA, Semigran MJ, Januzzi JL Jr. Heart failure outcomes and benefits of NT-proBNP-guided management in the elderly: results from the prospective, randomized ProBNP outpatient tailored chronic heart failure therapy (PROTECT) study. J Card Fail. 2012 Aug;18(8):626-34. doi: 10.1016/j.cardfail.2012.05.005. Epub 2012 Jun 19. PMID 22858078
- [Derived] Januzzi JL Jr, Rehman SU, Mohammed AA, Bhardwaj A, Barajas L, Barajas J, Kim HN, Baggish AL, Weiner RB, Chen-Tournoux A, Marshall JE, Moore SA, Carlson WD, Lewis GD, Shin J, Sullivan D, Parks K, Wang TJ, Gregory SA, Uthamalingam S, Semigran MJ. Use of amino-terminal pro-B-type natriuretic peptide to guide outpatient therapy of patients with chronic left ventricular systolic dysfunction. J Am Coll Cardiol. 2011 Oct 25;58(18):1881-9. doi: 10.1016/j.jacc.2011.03.072. PMID 22018299
- [Derived] Bhardwaj A, Rehman SU, Mohammed A, Baggish AL, Moore SA, Januzzi JL Jr. Design and methods of the Pro-B Type Natriuretic Peptide Outpatient Tailored Chronic Heart Failure Therapy (PROTECT) Study. Am Heart J. 2010 Apr;159(4):532-538.e1. doi: 10.1016/j.ahj.2010.01.005. PMID 20362709